CLINICAL TRIAL: NCT04223219
Title: Different Modalities of Analgesia in Open Heart Surgeries in Mansoura University: Randomized Prospective Comparative Study
Brief Title: Different Modalities of Analgesia in Open Heart Surgeries in Mansoura University
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Ahmed Gamal Morsy, Principle investigator, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD.19.11.255
Record Dates: First submitted 2019-12-28; First posted 2020-01-10 (Actual); Last update posted 2021-09-22 (Actual); Status verified 2021-09

CONDITIONS: Coronary Artery Disease; Valve Disease, Heart; Pain, Acute; Pain, Postoperative
MeSH Terms: conditions — Coronary Artery Disease; Heart Valve Diseases; Acute Pain; Pain, Postoperative | interventions — Fentanyl; Propofol; Dexmedetomidine; Ketamine; Magnesium Sulfate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: The study subjects will be blinded to the allocated groups. The outcome assessor (the investigator who will assess the primary and secondary outcomes) will be blinded to the allocated groups.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- High Opioid Group (Active Comparator): -The patients will receive fentanyl infusion at a rate of 1 µg/kg/h and fentanyl bolus 20-40 µg according to patient hemodynamics. (tachycardia: increase of heart rate >20% of baseline or hypertension: increase of mean blood pressure >20% of baseline).
  Interventions: Drug: Fentanyl
- Low Opioid Group (Placebo Comparator): The patients will receive fentanyl bolus 20 µg/hr and propofol 20 mg at the time of surgical stimulation and according to patient hemodynamics (repeated as required).
  Interventions: Drug: Fentanyl, Propofol
- Non-Opioid Group (Experimental): The patients will receive infusions of dexmedetomidine 0.2 µg/kg/h, ketamine 2 µg/kg/min, and magnesium sulfate 5 mg/kg/h.
  Interventions: Drug: Dexmedetomidine, Ketamine, Magnesium sulfate

INTERVENTIONS:
Drug: Fentanyl — * Induction of anesthesia : Midazolam 2 mg, Fentanyl 3 µg/kg, propofol 50-100 mg and Atracurium 0.5 mg/kg.
  * Maintenance of anesthesia (intraoperative until tracheal extubation):
  Maintenance will be achieved by isoflurane with concentration 0.5-1.5 % with 40% oxygen. During cardiopulmonary bypass by continuous infusion of Propofol at a rate of 2 mg/kg/hr. and Atracurium at a rate of 10 g/kg/min.
  * The patients will receive fentanyl infusion at a rate of 1 µg/kg/h and fentanyl bolus 20-40 µg according to patient hemodynamics. (tachycardia: increase of heart rate >20% of baseline or hypertension: increase of blood pressure >20% of baseline).
  * After tracheal extubation:
  all the patients will receive standard analgesia (i.v. paracetamol 1 gm every 12 hours and i.v. ketorolac 30 mg every 12 hours) and morphine patient controlled analgesia with bolus dose = 2 mg, lockout interval = 10 minutes, 4-hour dose limit = 10 mg, with no background infusion.
  Arms: High Opioid Group
Drug: Fentanyl, Propofol — * Induction of anesthesia : Midazolam 2 mg, Fentanyl 3 µg/kg, propofol 50-100 mg and Atracurium 0.5 mg/kg.
  * Maintenance of anesthesia (intraoperative until tracheal extubation):
  Maintenance of anesthesia will be achieved by isoflurane with concentration 0.5-1.5 % with 40% oxugen. During cardiopulmonary bypass by continuous infusion of Propofol at a rate of 2 mg/kg/hr. and Atracurium at a rate of 10 g/kg/min.
  * The patients will receive fentanyl bolus 20 µg/hr and propofol 20 mg at the time of surgical stimulation and according to patient hemodynamics (repeated as required).
  * After tracheal extubation:
  all the patients will receive standard analgesia (i.v. paracetamol 1 gm every 12 hours and i.v. ketorolac 30 mg every 12 hours) and morphine patient controlled analgesia with bolus dose = 2 mg, lockout interval = 10 minutes, 4-hour dose limit = 10 mg, with no background infusion.
  Arms: Low Opioid Group
Drug: Dexmedetomidine, Ketamine, Magnesium sulfate — * Induction of anesthesia : Midazolam 2 mg, Fentanyl 3 µg/kg, propofol 50-100 mg and Atracurium 0.5 mg/kg.
  * Maintenance of anesthesia (intraoperative until tracheal extubation):
  Maintenance of anesthesia will be achieved by isoflurane with concentration 0.5-1.5 % with 40% oxygen. During cardiopulmonary bypass by continuous infusion of Propofol at a rate of 2 mg/kg/hr. and Atracurium at a rate of 10 g/kg/min.
  * The patients will receive infusions of dexmedetomidine 0.2 µg/kg/h, ketamine 2 µg/kg/min, and magnesium sulfate 5 mg/kg/h.
  * After tracheal extubation:
  all the patients will receive standard analgesia (i.v. paracetamol 1 gm every 12 hours and i.v. ketorolac 30 mg every 12 hours) and morphine patient controlled analgesia with bolus dose = 2 mg, lockout interval = 10 minutes, 4-hour dose limit = 10 mg, with no background infusion.
  Arms: Non-Opioid Group

SUMMARY:
Cardiac surgery is associated with post-operative pain which is one of the major problems and remains one of the most controversial issues. Inadequate pain control after cardiac surgery increases the incidence of development of many complications. Intravenous opioids are commonly used for postoperative analgesia either on demand "physician or nurse-controlled" or patient -controlled.

Multimodal opioid sparing analgesia has become frequently used, These techniques can be achieved with Dexmedetomidine, low-dose ketamine and magnesium.

The study hypotheses that control of perioperative quality of pain with opioid sparing medications may improve analgesia and patient outcome.

DETAILED DESCRIPTION:
Pain after cardiac surgery is triggered by numerous factors including skin incision, sternotomy, sternal and rib retraction, internal mammary artery and saphenous vein harvesting, surgical manipulation of pleura, placement of chest tubes and tissue trauma during surgery.Median sternotomy significantly reduces postoperative pulmonary function; however, it is the most commonly used approach because it facilitates exposure of the surgical field.

Pain prevents early mobilization, reduction in pulmonary function and accumulation of bronchial secretions resulting in atelectasis, pulmonary infections, hypoxia and increase duration of ICU stay.Prolonged ICU stay is associated with greater risk of respiratory and renal dysfunction, and increases morbidity and mortality.

Optimal post-operative pain management allows early weaning from mechanical ventilation and extubation, early mobilization, facilitate beginning of chest physiotherapy, shortens the length of ICU stay and hospitalization, medical costs and decreases incidence of post-operative complications.

Opioid infusions and patient-controlled analgesia (PCA) remain the principal and most commonly used for immediate postoperative analgesia after cardiac surgery in Intensive Care Units.

Multimodal opioid sparing analgesia has become frequently used. They are used for the opioids sparing effect and for achievement of a more efficient pain management via both central and peripheral anti-nociceptive mechanisms.

Dexmedetomidine is an intravenous α-2 agonist widely used for sedation, anxiolysis and for augmenting anesthesia and analgesia with reduction in opioid requirements. Ketamine have a great analgesic effect and can be added to multimodal regimen. Magnesium can be added to multimodal regimen as it acts as a non-competitive antagonist of N-methyl-D-aspartate (NMDA) receptors and has anti-inflammatory effects and can be used in acute pain management.

The aim of this study is to compare between traditional high opioid, low opioid and non-opioid technique on the patient outcome.

This prospective randomized comparative study will be conducted on 75 patients undergoing cardiac procedures that will require cardiopulmonary bypass and median sternotomy at Cardiothoracic Surgical Department, Mansoura University Hospitals over 24 months.

Eligible 90 patients will be randomly allocated to one of three equal groups each contains 25 patients, they will be randomized according to computer-generated randomization sequence: Either high opioid group (group I), Low opioid group (group II) and non-opioid group (group III).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of both gender,
* Aged above 18 years
* American Society of Anesthesiologists (ASA) physical status II & III,
* Body mass index less than 40 kg/m2
* Scheduled for any cardiac procedure with median sternotomy that require cardiopulmonary bypass at Cardiothoracic Surgical Department, Mansoura University Hospitals.

Exclusion Criteria:

* Patients with pulmonary dysfunction or chronic obstructive pulmonary diseases
* Acute or unstable angina
* Previous cardio-thoracic surgery
* Emergency surgery
* Left ventricular ejection fraction less than 40%
* Dysrhythmia or pacemaker
* Major hepatic or renal dysfunction
* Need for re-exploration, uncontrolled diabetes (HbA1c > 8.5)
* Neurological deficit
* Hyper-magnesemia

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2019-12-10 (Actual); Primary Completion 2021-08-15 (Actual); Study Completion 2021-09-15 (Estimated)

PRIMARY OUTCOMES:
Pain score at rest assessed using the visual analogue scale. | 30 minutes after tracheal extubation
  visual analogue scale is a straight horizontal line of fixed length, usually 100 mm. orientated from the left (worst) to the right (best) (where 0 is no pain and 100 is the worst pain) lower score means better outcome

SECONDARY OUTCOMES:
Pain score at rest assessed using the visual analogue scale. | 2, 6, 12, and 24 hours after tracheal extubation
  visual analogue scale is a straight horizontal line of fixed length, usually 100 mm. orientated from the left (worst) to the right (best) (where 0 is no pain and 100 is the worst pain) lower score means better outcome
Sedation level assessed using Ramsay sedation score | 30 minutes, 2, 6, 12, and 24 hours after tracheal extubation
  Ramsay sedation score used to assess level of sedation range from 1 to 6 where (1: awake, anxious, agitated, restless, 2: awake, cooperative, orientated, and tranquil, 3: responsive to commands only, 4: asleep, brisk response to light glabellar tap or loud auditory stimulus, 5: asleep, sluggish response to light glabellar tap or loud auditory stimulus and, 6: no response to light glabellar tap or loud auditory stimulus).
  lower score means better outcome
Heart rate | every 15 minutes in the first hour then every 30 minutes intraoperative and then 1 hour post-operative
Systolic blood pressure | every 15 minutes in the first hour then every 30 minutes intraoperative and then 1 hour post-operative
Diastolic blood pressure | every 15 minutes in the first hour then every 30 minutes intraoperative and then 1 hour post-operative
Mean arterial blood pressure | every 15 minutes in the first hour then every 30 minutes intraoperative and then 1 hour post-operative
Total opioid consumption | 24 hours post operative
  calculation of total opioids used intra operative and pos operative
Time to tracheal extubation | 2 hours to 6 hours
Duration of ICU stay | 2 to 5 days
Time to either bowel movement or flatus | within 24 hours
Number of participants with post-operative nausea and vomiting (PONV) | within 24 hours
Doses of atropine required | from start to the end of surgery
Doses of Inotropic required | from start to the end of surgery
Doses of vasopressors required | from start to the end of surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura Faculty of medicine, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Undecided